#### Cover Page for Clinical Trials Document posting

Official Title: S1400F, "A Phase II Study of MEDI4736 (Durvalumab) Plus Tremelimumab as Therapy

for Patients with Previously Treated Anti-PD-1/PD-L1 Resistant Stage IV Squamous Cell

Lung Cancer (Lung-MAP Non-Match Sub-Study)"

NCT Number: 03373760

Version Date: 10/21/2019

Description:

**\$1400** [NCT 02154490] is the parent study to **\$1400F** [NCT 03373760].

The **<u>\$1400</u>** Lung-MAP study is considered one study under one IND consisting of:

• S1400 Version Control Protocol

- S1400 Main Screening Protocol Component
- Multiple Sub-Studies (or sub-protocols) Components

Each component is contained in its own separate document.

<u>S1400F</u> is one of these components. Each "component" consists of the protocol document and its associated informed consent document(s). Since each screening and sub-study component operates independently from the other components contained in Lung-MAP, each has its own version date and NCT number. This is due to the complexity of the study and how it must be entered into different computer programs.

## **Informed Consent Model for S1400F**

## \*NOTES FOR LOCAL INSTITUTION INFORMED CONSENT AUTHORS:

This model informed consent form has been reviewed by the DCTD/NCI and is the official consent document for this study. Local IRB changes to this document are allowed. (Institutions should attempt to use sections of this document that are in bold type in their entirety.) Editorial changes to these sections may be made as long as they do not change information or intent. If the institutional IRB insists on making additions, deletions, or more substantive modifications to the risks or alternatives sections, they may be justified in writing by the investigator and approved by the IRB. Under these circumstances, the revised language, justification and a copy of the IRB minutes must be forwarded to the SWOG Operations Office for approval before a patient may be registered to this study.

Please particularly note that the questions related to banking of specimens for future study are in bolded type and may not be changed in any way without prior approval from the SWOG Operations Office.

| Readability Statistics: | | |
|----------------------------|------|----------------------|
| Flesch Reading Ease | 61.5 | (targeted above 55) |
| Flesch-Kincaid Grade Level | 8.7 | (targeted below 8.5) |

- Instructions and examples for informed consent authors are in [italics].
- A blank line, \_\_\_\_\_\_, indicates that the local investigator should provide the appropriate information before the document is reviewed with the prospective research participant.
- The term "study doctor" has been used throughout the model because the local investigator for a cancer treatment trial is a physician. If this model is used for a trial in which the local investigator is not a physician, another appropriate term should be used instead of "study doctor".
- The dates of protocol updates in the header and in the text of the consent is for reference to this model only and should not be included in the informed consent form given to the prospective research participant.
- The local informed consent must state which parties may inspect the research records. This includes the NCI, the drug manufacturer for investigational studies, any companies or grantors that are providing study support (these will be listed in the protocol's model informed consent form) and SWOG.
- "SWOG" must be listed as one of the parties that may inspect the research records in all protocol consent forms for which patient registration is being credited to SWOG. This includes consent forms for studies where all patients are registered directly through the SWOG Data Operations Office, all intergroup studies for which the registration is being credited to SWOG (whether the registration is through the SWOG Data Operations



Office or directly through the other group), as well as consent forms for studies where patients are registered via CTSU and the registration is credited to SWOG

• When changes to the protocol require revision of the informed consent document, the IRB should have a system that identifies the revised consent document, in order to preclude continued use of the older version and to identify file copies. An appropriate method to identify the current version of the consent is for the IRB to stamp the final copy of the consent document with the approval date. The stamped consent document is then photocopied for use. Other systems of identifying the current version of the consent such as adding a version or approval date are allowed as long as it is possible to determine during an audit that the patient signed the most current version of the consent form.

#### \*NOTES FOR LOCAL INVESTIGATORS:

- The goal of the informed consent process is to provide people with sufficient information for making informed choices. The informed consent form provides a summary of the clinical study and the individual's rights as a research participant. It serves as a starting point for the necessary exchange of information between the investigator and potential research participant. This model for the informed consent form is only one part of the larger process of informed consent. For more information about informed consent, review the "Recommendations for the Development of Informed Consent Documents for Cancer Clinical Trials" prepared by the Comprehensive Working Group on Informed Consent in Cancer Clinical Trials for the National Cancer Institute. The Web site address for this document is http://cancer.gov/clinicaltrials/understanding/simplification-of-informed-consent-docs/
- A blank line, \_\_\_\_\_, indicates that the local investigator should provide the appropriate information before the document is reviewed with the prospective research participant.
- Suggestion for Local Investigators: An NCI pamphlet explaining clinical trials is available for your patients. The pamphlet is titled: "Taking Part in Cancer Treatment Research Studies". This pamphlet may be ordered on the NCI Web site at <a href="https://cissecure.nci.nih.gov/ncipubs">https://cissecure.nci.nih.gov/ncipubs</a> or call 1-800-4- CANCER (1-800-422-6237) to request a free copy.
- Optional feature for Local Investigators: Reference and attach drug sheets, pharmaceutical information for the public, or other material on risks. Check with your local IRB regarding review of additional materials.

\*These notes for authors and investigators are instructional and should not be included in the informed consent form given to the prospective research participant.



# Study Title for Study Participants: Targeted Treatment for Advanced Squamous Cell Lung Cancer

## Official Study Title for Internet Search on

http://www.ClinicalTrials.gov:

<u>S1400</u>, "A Biomarker-Driven Master Protocol for Previously Treated Squamous Cell Lung Cancer"

<u>LUNGMAP</u>, "A Master Protocol to Evaluate Biomarker-Driven Therapies and Immunotherapies in Previously-Treated Non-Small Cell Lung Cancer"

<u>S1400F</u>, "A Phase II Study of MEDI4736 (Durvalumab) plus Tremelimumab as Therapy for Patients with Previously Treated ANTI-PD-1/PD-L1 Resistant Stage IV Squamous Cell Lung Cancer (Lung-MAP Non-Match Sub-Study)"

## What is the usual approach to my lung cancer?

You are being asked to take part in this study because you have squamous cell lung cancer. Various chemotherapy drugs have been shown to improve survival for patients with advanced squamous lung cancer. People who are not on this study are usually treated at first with cisplatin or carboplatin in combination with a second chemotherapy drug such as gemcitabine, paclitaxel, docetaxel, or vinorelbine. In addition, immunotherapy drugs called nivolumab and pembrolizumab were recently FDA approved for patients with squamous lung cancer who previously received chemotherapy.

## What are my other choices if I do not take part in this study?

Your other choices may include:

- You may choose to have the usual approach described above
- You may choose to take part in a different study, if one is available
- You may choose to get comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

## Why is this study being done?

There are several investigational treatments that are being tested in various sub-studies as part of this study. You will have already received the information on your biomarker testing. You have been assigned to this treatment study because you did not have a biomarker match and received immunotherapy as your most recent treatment. For this sub-study, you will be given two



treatments, MEDI4736 and tremelimumab, a treatment that is designed to help your immune system fight the cancer. The purpose of this sub-study is to look at the effects (good and bad) of MEDI4736 combined with tremelimumab. MEDI4736 and tremelimumab are investigational for this study. MEDI4736 and tremelimumab may or may not shrink your cancer and they could cause side effects.

We expect about 132 patients to be registered to this sub-study.

## What are the study groups?

You have been assigned to this sub-study because your tumor sample did not have any of the biomarkers being tested in the other sub-studies or you were not eligible to participate in the other sub-studies. This sub-study is a single arm study with two groups. Each group will receive the same treatment. The first group are patients with no change in their tumor growth 24 weeks after starting immunotherapy. The second group are patients with tumor growth within 24 weeks of starting immunotherapy.

Tremelimumab will be given through your vein over 60 minutes followed by a 60 minute observation time before you are then given MEDI4736 through your vein over 60 minutes. If the infusion is well tolerated, the observation period may be reduced from one hour at the study doctor's discretion. A cycle is 28 days. MEDI4736 and Tremelimumab will be given on Day 1 of Cycles 1, 2, 3 and 4. MEDI4736 will be given alone on Day 1 of Cycle 5 and subsequent cycles.

The treatment on this study is described in the table below.

| Drug | How often is it given? | How is it given? | What days is it given on? | What is the cycle duration? |
|---|---|---|---|---|
| Tremelimumab | Once, every<br>28 days (up to<br>4 doses) | Into a vein over 60 minutes | Day 1 of<br>Cycle 1-4 | 28 days |
| MEDI4736 | Once, every<br>28 days | Into a vein over 60 minutes | Day 1 | 28 days |

Another way to find out what may happen to you during the study is to read the chart below. Start reading at the top of the chart and read down, following the arrows.





## How long will I be in this study?

The total amount of time you will take part in this research study will depend on how your cancer is responding to the study treatment. After you are finished receiving study treatment, the study doctor will continue to watch you for side effects and follow your condition every 3 months for the first year, then every 6 months up to three years from the time you started treatment. The study doctor will ask you to visit the office for follow up physical exams, blood tests, and scans. Your doctor may give you other tests or procedures if they think they are needed for the regular care of your disease.

## What extra tests and procedures will I have if I take part in this study?

Most of the exams, tests, and procedures you will have are part of the usual approach for your cancer. However, there are some extra exams, tests, and/or procedures that you will need to have if you take part in this study.

The leftover tumor sample from the screening biomarker testing will undergo an additional lab test. The test is being performed to see if you have a biomarker call PD-L1. PD-L1 is a genetic feature or specific protein found in the tumor sample. You will not have another surgery. The samples will be kept until there are no additional sub-studies for you to enroll in or they are used up, whichever happens first. If any tumor is left over after the laboratory studies and there are no additional sub-studies for you to enroll in, and if you agreed, it will be stored for biobanking. This was discussed in the screening consent section on optional studies.

#### Before you begin the study:

You will need to have the following extra test to find out if you can be in the study:

• Blood test to assess the levels of hormones coming from your thyroid.

If the exams, tests, and procedures show that you can take part in the study, and you choose to take part, then you will need the following extra test.



During the study:

• Blood test to assess the function of the thyroid gland levels of hormones coming from your thyroid

The blood test will be repeated approximately on Day 1 of every cycle while you are receiving treatment, then only as needed until your disease worsens.

Neither you nor your health care plan/insurance carrier will be billed for the thyroid tests that will be used for this study.

## What possible risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that the treatment may not be as good as the usual approach for your cancer or condition at shrinking or stabilizing your cancer.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The treatment used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drug(s)/study approach.

Here are important things to know about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, and some may never go away.
- Some side effects may make it hard for you to have children.
- Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

The tables below show the most common and the most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.



#### Possible Side Effects of MEDI4736

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving MEDI4736 (durvalumab), more than 20 and up to 100 may have:

• Cough

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving MEDI4736 (durvalumab), from 4 to 20 may have:

- Pain in the muscles, joints
- Diarrhea, nausea, vomiting
- Swelling of the body
- Tiredness, fever
- Infections. Infections can be severe and involve jaws and fatty tissues
- Loss of appetite
- Painful urination
- Shortness of breath
- Change in voice
- Increased sweating

MEDI4736 (durvalumab) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Hormone gland problems (especially the thyroid, pituitary and adrenal glands). Signs and symptoms may include: headaches, extreme tiredness or changes in mood or behavior; decreased sex drive; weight loss or weight gain; excessive thirst or urine; dizziness or fainting
- Liver problems (hepatitis) which can cause liver failure. Signs and symptoms of hepatitis may include: yellowing of your skin or the whites of your eyes, severe nausea or vomiting; drowsiness; pain in the right upper belly
- Lung problems (including pneumonitis), symptoms may include: new or worsening cough, chest pain, shortness of breath
- Skin: itching; rash; patches of light skin color

#### RARE, AND SERIOUS

In 100 people receiving MEDI4736 (durvalumab), 3 or fewer may have:

• Reaction during or after infusion which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat



MEDI4736 (durvalumab) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Damage to blood cells that may cause bruises and bleeding
- Blood clots in small blood vessels, which may cause kidney failure, fever, and confusion
- Heart problems including heart failure. Symptoms and signs of heart problems may include: shortness of breath, swelling of the ankle and body or abnormal heartbeat
- A condition with high blood sugar (diabetes) which leads to tiredness, frequent urination or excessive thirst which may require treatment with insulin
- Swelling and redness of the eye
- Intestinal problems (colitis) that can rarely lead to tears or holes in your intestine. Signs and symptoms may include: diarrhea or increase in bowel movements, belly pain, bloody or dark, tarry, sticky stools
- Damage to the pancreas which may cause belly pain and hospitalization
- Problem of the muscle (myositis), which can cause muscle pain and severe muscle weakness sometimes with dark urine
- Swelling of the brain, which may cause headache, blurred vision, stiff neck, and/or confusion
- Problem of the nervous system that can cause weakness and paralysis, which may include: numbness, tingling of hands and feet, and may also cause problems with breathing
- Kidney problems, including kidney failure requiring dialysis. Signs of kidney problems may include: decrease in the amount of urine, blood in your urine, ankle swelling
- Severe skin reactions with blisters and peeling which can involve mouth and other parts of the body

### **Possible Side Effects of Tremelimumab**

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving tremelimumab, more than 20 and up to 100 may have:

• Diarrhea

Tremelimumab (CP-675, 206) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

• Skin: itching; dry; rash (may be raised); skin change; hives



## OCCASIONAL, SOME MAY BE SERIOUS In 100 people receiving tremelimumab, from 4 to 20 may have:

- Swelling and redness of the eye
- Belly pain
- Nausea, vomiting
- Swelling of arms, legs
- Tiredness, fever
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Bruising, bleeding
- Infection, especially when white blood cell count is low
- Loss of appetite, dehydration
- Cough, shortness of breath

Tremelimumab (CP-675, 206) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Anemia which may require blood transfusion
- Hormone gland problems (especially the thyroid, pituitary and adrenal glands, and pancreas). Signs and symptoms may include: headaches that will not go away or unusual headaches, extreme tiredness or changes in mood or behavior; decreased sex drive; weight loss or weight gain; excessive thirst or urine; dizziness or fainting.
- Intestinal problems (colitis) that can rarely lead to tears or holes in your intestine and
  may require surgery. Signs and symptoms of colitis may include: diarrhea or increase
  in bowel movements, blood in your stools or dark, tarry, sticky stools, severe belly
  pain or tenderness
- Pain or swelling of joints
- Problem of the muscle, including swelling, which can cause muscle pain and severe muscle weakness sometimes with dark urine
- Problem of the nerves that can cause paralysis. Signs and symptoms may include: numbness, tingling of hands and feet; weakness of the arms, legs and facial muscle movement.
- Lung problems (pneumonitis). Symptoms may include: new or worsening cough, chest pain, shortness of breath.
- Kidney damage which may cause swelling, may require dialysis



## RARE, AND SERIOUS In 100 people receiving tremelimumab (CP-675, 206), 3 or fewer may have:

- Damage to the heart
- A condition with high blood sugar which leads to tiredness, frequent urination or excessive thirst
- Dry mouth and dry eyes which may become permanent
- Damage to the skin which may cause tightening and abnormal movement of arms and legs

Tremelimumab (CP-675, 206) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Swelling of the bowels
- Damage to the pancreas which may cause belly pain and hospitalization
- Liver problems (hepatitis) which can cause liver failure. Signs and symptoms of hepatitis may include: yellowing of your skin or the whites of your eyes, severe nausea or vomiting; drowsiness; pain in the right upper belly
- Swelling of the brain (encephalitis), which may cause: headache, confusion, sleepiness, seizures, and stiff neck
- Swelling of the blood vessels of the scalp which may become severe and may be lifethreating

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

Reproductive risks: You should not get pregnant, breastfeed, or father a baby while in this study as the drugs used in this study could be very damaging to an unborn baby. Women who receive study drug should use effective contraception during the period of the trial and for at least 180 days after completion of treatment. Check with the study doctor about what types of birth control, or pregnancy prevention, to use while in this study.

## What possible benefits can I expect from taking part in this study?

It is not possible to know at this time if the study drug/study approach is better than the usual approach, so this study may or may not help you. This study will help researchers learn things that will help people in the future.

## Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide



whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- If you do not follow the study rules
- If the study is stopped by the sponsor, IRB or FDA.

## What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

| For questions about your rights while in this study, call the | |
|---|---|
| (insert name of center) Institutional Review Board at | (insert telephone |
| number). (Note to Local Investigator: Contact information for patient repre | esentatives or other |
| individuals at a local institution who are not on the IRB or research team b | ut take calls |
| regarding clinical trial questions can also be listed here.) | |

## What are the costs of taking part in this study?

The MEDI4736 and tremelimumab will be supplied at no charge while you take part in this study. The cost of getting MEDI4736 and tremelimumab ready and giving it to you is not paid by the study sponsor so you or your insurance company may have to pay for this. It is possible that the MEDI4736 and tremelimumab may not continue to be supplied while you are on the study. Although not likely, if this occurs, your study doctor will talk to you about your options.

You and/or your health plan/insurance company will need to pay for all of the other costs of treating your cancer while in this study, including the cost of tests, procedures, or medicines to manage any side effects, unless you are told that certain tests are supplied at no charge. Before you decide to be in the study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will not be paid for taking part in this study.

## What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for



injury. Your insurance company may not be willing to pay for study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a study.

### Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The study sponsor, SWOG, and the drug company supporting the treatment sub-study you are on.
- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration (FDA) and the National Cancer Institute (NCI) in the U.S., and similar ones if other countries are involved in the study.
- Transmission of Imaging and Data (TRIAD) and Imaging and Radiation Oncology Core (IROC)-Your medical images with clinical study data (e.g., the treatment Group you are assigned to, etc.) will be transferred via TRIAD to IROC at Ohio State University in Columbus, Ohio. Your medical images will be reviewed by physicians at this organization as part of the study analysis for this trial. In addition, information gained from this study may be used in the future for additional research and only that data would be provided to other scientist for future research. Your name, and any other information that could be used to identify you personally, will not be included.

## Where can I get more information?

You may visit the NCI Web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.



## Who can answer my questions about this study?

| You can talk to the study of | loctor about any questions or concerns ye | ou have about this study or to |
|---|---|---|
| report side effects or injuri | es. Contact the study doctor | (insert name of |
| study doctor[s]) at | (insert telephone number | r). |

#### **OPTIONAL STUDIES SECTION**

## This section is about optional studies you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. You will not get health benefits from any of these studies. The researchers leading this optional study hope the results will help other people with cancer in the future.

The results will not be added to your medical records, nor will you or your study doctor know the results.

You will not be billed for these optional studies. You can still take part in the main study even if you say 'no' to any or all of these studies. If you sign up for but cannot complete any of the studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for each of the following studies.

## 1. Optional Additional Biopsy and Optional Sample Collections for Laboratory Studies and/or Biobanking for Possible Future Studies

Researchers are trying to learn more about cancer, diabetes, and other health problems. Much of this research is done using samples from your tissue, blood, urine, or other fluids. Through these studies, researchers hope to find new ways to prevent, detect, treat, or cure health problems.

Some of these studies may be about genes. Genes carry information about features that are found in you and in people who are related to you. Researchers are interested in the way that genes affect how your body responds to treatment.

If you choose to take part, tissue and blood specimens will be collected in this part of the study and the researchers would like to ask your permission to store and use your samples and health information for medical research. The research that may be done is unknown at this time. Storing samples for future studies is called "biobanking". The Biobank is being run by SWOG and supported by the National Cancer Institute.

#### WHAT IS INVOLVED?

If you agree to take part, here is what will happen next:

1) Your specimens may be stored in the Biobank, along with samples from other people who take part. These specimens may include:



- About 2 tablespoons of blood will be collected from a vein in your arm (at the same time as other study blood tests) before the study and on Weeks 5, 9, and 13.
  - The most common risks related to drawing blood from your arm are brief pain and possibly a bruise.
- A sample of tissue will be collected from an optional extra biopsy before starting treatment on this study. If you provided a fresh biopsy during your biomarker testing and received no additional treatment, that leftover tissue may be used for this optional biopsy.
- A sample of tissue will be collected from an optional extra biopsy after treatment if your cancer gets worse on this study.
  - Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, pain and bruising at the biopsy site, which can be treated with regular pain medications. Rarely, an infection can occur. You will sign a separate consent form before the biopsy is taken. This will be a standard surgical consent form from the institution where the biopsy procedure takes place. Rarely, patients may experience partial lung collapse that may require a chest tube or even a breathing machine. The samples will be kept until they are used up.
- Qualified researchers can submit a request to use the materials stored in the Biobanks. A science committee at the clinical trials organization, and/or the National Cancer Institute, will review each request. There will also be an ethics review to ensure that the request is necessary and proper. Researchers will not be given your name or any other information that could directly identify you.
- 3) Neither you nor your study doctor will be notified when research will be conducted or given reports or other information about any research that is done using your samples.
- 4) Some of your genetic and health information may be placed in central databases that may be public, along with information from many other people. Information that could directly identify you will not be included.

#### WHAT ARE THE POSSIBLE RISKS?

- 1) There is a risk that someone could get access to the personal information in your medical records or other information researchers have stored about you.
- 2) There is a risk that someone could trace the information in a central database back to you. Even without your name or other identifiers, your genetic information is unique to you. The researchers believe the chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information.
- 3) In some cases, this information could be used to make it harder for you to get or keep a job or insurance. There are laws against the misuse of genetic information, but they may not give full protection. There can also be a risk in knowing genetic information. The Genetic Information Nondiscrimination Act of 2008, also referred to as GINA,



was passed by Congress to protect Americans from such discrimination. The law prevents discrimination from health insurers and employers. This law does not cover life insurance, disability insurance and long-term care insurance. New health information about inherited traits that might affect you or your blood relatives could be found during a study. The researchers believe the chance these things will happen is very small but cannot promise that they will not occur.

### HOW WILL INFORMATION ABOUT ME BE KEPT PRIVATE?

Your privacy is very important to the researchers and they will make every effort to protect it. Here are just a few of the steps they will take:

- 1) When your samples are sent to the researchers, no information identifying you (such as your name) will be sent. Samples will be identified by a unique code only.
- 2) The list that links the unique code to your name will be kept separate from your sample and health information. Any Biobank and SWOG staff with access to the list must sign an agreement to keep your identity confidential.
- 3) Researchers to whom SWOG sends your sample and information will not know who you are. They must also sign an agreement that they will not try to find out who you are.
- 4) Information that identifies you will not be given to anyone, unless required by law.
- 5) If research results are published, your name and other personal information will not be used.

### WHAT ARE THE POSSIBLE BENEFITS?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

#### ARE THERE ANY COSTS OR PAYMENTS?

Neither you nor your health care plan/insurance carrier will be billed for the collection or testing of the tumor tissue or blood samples that will be used for this study. You will not be paid for taking part. If any of the research leads to new tests, drugs, or other commercial products, you will not share in any profits.

#### WHAT IF I CHANGE MY MIND?

| If you decide you no longer want your samples to be used, you can call the study doctor, |
|---|
| , (insert name of study doctor for main trial) at |
| (insert telephone number of study doctor for main trial) who will let the researchers know. Then |
| any sample that remains in the bank will no longer be used. |

Samples or related information that have already been given to or used by researchers will not be returned.



## WHAT IF I HAVE MORE QUESTIONS?

| If you | - | at the use of your samples for research, contact the study doctor,<br>rt name of study doctor for main trial), at |
|---|---|---|
| (inser | | of study doctor for main trial). |
| Pleas | e circle your answer | to show whether or not you would like to take part in each option: |
| SAN | IPLES FOR FUT | TURE RESEARCH STUDIES: |
| 1. | I agree to have an<br>treatment on this<br>YES | optional biopsy to collect a sample of tissue before starting study. NO |
| 2. | If my cancer responds to study treatment, I agree to have another biopsy after completing study treatment to collect a sample of tissue. YES NO | |
| 3. | My tumor tissue a health research. | and related information may be kept in a Biobank for use in future |
| | YES | NO |
| 4. | My blood samples and related information may be kept in a Biobank for use if future health research. | |
| | YES | NO |
| This | is the end of the secti | on about optional studies. |
| My S | Signature Agreei | ng to Take Part in the Main Study |
| my qı | uestions have been ar | rm, or had it read to me. I have discussed it with the study doctor and aswered. I will be given a signed copy of this form. I agree to take part additional studies where I circled 'yes'. |
| Partic | cipant's signature | |
| Date | of signature | |
| | | and date lines for the person(s) conducting the discussion may be of the study sponsor.) |
| Signa | ature of person(s) con | ducting the informed consent discussion |
| Date | of signature | |



## Informed Consent Addendum Model for <u>S1400F</u> at Progression for Continued Treatment

<u>S1400</u>, "A Biomarker-Driven Master Protocol for Previously Treated Squamous Cell Lung Cancer"

<u>LUNGMAP</u>, "A Master Protocol to Evaluate Biomarker-Driven Therapies and Immunotherapies in Previously-Treated Non-Small Cell Lung Cancer"

<u>S1400F</u>, "A Phase II Study of MEDI4736 (Durvalumab) plus Tremelimumab as Therapy for Patients with Previously Treated ANTI-PD-1/PD-L1 Resistant Stage IV Squamous Cell Lung Cancer (Lung-MAP Non-Match Sub-Study)"

The following information should be read as an update to the original Consent form that you read and signed at the beginning of the study. Unless specifically stated otherwise in the following paragraphs, all information contained in that original Consent Form is still true and remains in effect. Your participation continues to be voluntary. You may refuse to participate or may withdraw your consent to participate at any time, and for any reason, without jeopardizing your future care at this institution or your relationship with your study doctor.

At this point in your care, your cancer has grown, so you are being asked whether you want to stay on this study and continue receiving study treatment, or whether you want to stop taking study treatment.

The usual approach to treating people whose cancer has grown on a standard treatment (not study treatment) is usually to continue with the same treatment while it is still providing clinical benefit or to get treated with chemotherapy such as docetaxel (or other drugs). Clinical benefit means that your treatment has shown a positive effect on how you feel, and that you continue to feel well on treatment even though your scans show cancer growth.

Other choices if you do not choose to continue receiving treatment on this study are:

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

By signing below, you are stating that you and your study doctor have talked about your options and have decided to continue receiving study treatment as it is providing clinical benefit.



### **Patient Signature and Date**

By signing this form, I acknowledge that I have read the information above or had it read to me. I have discussed it with a member of the study team and my questions have been answered. I understand that I will be given a copy of this form.

| Participant's signature |
|-------------------------|
| Date of signature |

